CLINICAL TRIAL: NCT06999031
Title: An Exploratory Clinical Study on the Safety and Efficacy of Autologous T Cell Injection Targeting BCMA Chimeric Antigen Receptor (CG-105-12) in the Treatment of Patients With Relapsed / Refractory Multiple Myeloma
Brief Title: A Study to Evaluate CG-105-12 in Patients With Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Collaborators: Cells & Genes Biotech (Shanghai) Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-105-12
Record Dates: First submitted 2025-05-15; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Relapsed/Refractory; Multiple Myeloma
Keywords: multiple myeloma; relapsed/refractory; chimeric antigen receptor T Cell; BCMA
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group CG-105-12 (Experimental): Biological: BCMA-Targeted Chimeric Antigen Receptor Autologous T-cell
  Interventions: Biological: BCMA-Targeted Chimeric Antigen Receptor Autologous T-cell

INTERVENTIONS:
Biological: BCMA-Targeted Chimeric Antigen Receptor Autologous T-cell — Chimeric Antigen Receptor Autologous T-cell

SUMMARY:
This study is a single-centre, single-arm, open-label, dose-escalation exploratory study with single-dose administration. Its objective is to evaluate the safety, tolerability, dose, anti-tumor efficacy, and pharmacokinetic characteristics of CG-105-12 in the participants with BCMA-positive relapsed/refractory multiple myeloma who previously received adequate but uneffective standard treatments.

DETAILED DESCRIPTION:
This study is a single-centre, open-label, dose-escalation exploratory clinical trial. Its objective is to evaluate the safety, tolerability, recommended dose, anti-tumor efficacy, and pharmacokinetic characteristics of CG-105-12 infused in participants with BCMA-positive relapsed/refractory multiple myeloma who previously received adequate but uneffective standard treatments.. The study will be carried out in accordance with the protocol. Due to the early-stage of the exploratory clinical research,, the anticipated sample size for the three dose groups is 7-12 participants.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 18-75 years (inclusive of 18 and 75 years old), gender not limited;
* 2.Subject has received at least 3 lines of therapy, including at least proteasome inhibitors (PIs) and immunomodulatory therapy (IMiD); disease relapse, progression, or refractory according to the International Myeloma Working Group (IMWG) Consensus (2016) criteria for multiple myeloma;
* 3.Subjects whose tumor specimens were positive for BCMA expression on the membrane surface of plasma cells by immunohistochemistry (IHC) or flow cytometry and had not received prior BCMA CAR-T therapy;
* 4.One of the following is met (all data below are compared to the obtained minimum values):
* - a. Serum M-protein increased by more than 25% (absolute increase greater than 5 g/L) or M-protein increased by more than 10 g/L (if baseline serum M-protein is greater than 50 g/L);
* - b. Uroprotein increased by more than 25% (absolute increase greater than 200 mg/24h);
* - c. The difference between affected and unaffected serum FLC increased by more than 25% and the absolute value increased by more than 100 mg/L;
* - d.The proportion of bone marrow plasma cells increased by more than 25% and the absolute value increased by more than 10%;
* - e. The sum of the original maximum vertical diameter products of more than one measurable lesion increased by at least 50% from the lowest point; or the long axis of the original lesion of at least 1 cm increased by at least 50%;
* - f. An increase in circulating plasma cells of at least 50% (used when only circulating plasma cells are measurable lesions, with an absolute value of at least 200 cells per microlitre);
* 5.ECOG performance status score of 0-2；
* 6.Expected survival ≥12 weeks；
* 7.Subjects must have adequate organ function and meet all of the following laboratory test results prior to enrollment:
* - a.Complete blood count: Neutrophil count (ANC) 1E9/L; Lymphocyte count (ALC) 0.5E9/L; Platelet count >50E9/L; Haemoglobin >60g/L or Haematocrit >0.24；
* - b.Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 2.5 times the upper limit of normal (ULN); serum total bilirubin less than 1.5 times the ULN;
* - c.Renal function: The creatinine clearance rate calculated according to the Cockcroft-Gault formula is GFR 40ml/min (except for those whose renal function is abnormal due to progression of the primary disease as judged by the investigator);
* - d.Coagulation function: fibrinogen ≥ 1.0 g/L; activated partial thromboplastin time ≤1.5×ULN, prothrombin time (PT) ≤ 1.5×ULN;
* - e.Blood oxygen saturation > 91%;
* - f.Left ventricular ejection fraction (LVEF) ≥ 50%;
* 8.Subjects and their spouses agreed to use effective instrumental or medical contraception (except for safe contraception) from the time of signing the informed consent form until one year after CAR-T cell reinfusion;
* 9.Participants must personally sign a written informed consent form approved by the Ethics Committee prior to the start of any screening procedure.

Exclusion Criteria:

* 1.Hepatitis B surface antigen (HBsAg) positive, or Hepatitis B core antibody (HBcAb) positive with detectable Hepatitis B Virus (HBV) DNA in peripheral blood; Hepatitis C Virus (HCV) antibody positive with peripheral blood positive for Hepatitis C Virus (HCV) RNA; Human Immunodeficiency Virus (HIV) antibody positive; and Syphilis test positive.
* 2.Prior antitumor therapy as follows:
* - a.Treatment of multiple myeloma with monoclonal antibodies, CNS radiotherapy within 8 weeks prior to single nucleated cell collection;
* - b.or cytotoxic chemotherapy, immunomodulator therapy, or proteasome inhibitor therapy within 14 days prior to single nucleated cell collection;
* - c.or have received granulocyte-macrophage colony-stimulating factor (GM-CSF), long-acting granulocyte colony-stimulating factor (G-CSF) within 14 days prior to the single nucleated cell collection;
* 3.Has used therapeutic doses of corticosteroids (defined as prednisone or equivalent >20 mg/day) within 7 days prior to screening, but physiologic replacement, topical and inhaled steroids are permitted;
* 4.have received treatment containing bendamustine or fludarabine within 12 weeks prior to screening;
* 5.Plasma cell leukemia, patients suspected or suspected of having plasma cell tumor central nervous system invasion during screening;
* 6.patients with previous allogeneic hematopoietic stem cell transplantation;
* 7.malignancies other than multiple myeloma within 5 years prior to screening, excluding adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancers, localized prostate cancer after radical surgery, and ductal carcinoma in situ of the breast after radical surgery;
* 8.subjects with a history of solid organ transplantation;
* 9.Subjects who have undergone major surgery ( 3 level) within 2 weeks prior to the collection of individual nuclear cells, or who plan to have surgery within 2 weeks after the study treatment (subjects who plan to have local anesthesia surgery can participate in this study);
* 10.have received a live attenuated vaccine within ≤ 4 weeks prior to administration of the pretreatment regimen;
* 11.Presence of severe underlying diseases, such as:
* - a.Patients with autoimmune diseases (systemic lupus erythem- atosus, multiple sclerosis, rheumatoid arthritis, etc.) who need long-term use of immunosuppressants (methotrexate, cycl - ophosphamide, etc.), biological agents (infliximab, tozumab, etc.), glucocorticoids (prednisone, dexamethasone, etc.);
* - b.Uncontrolled active infection within 7 days prior to collection of a single nuclear cell, and evidence of severe active viral, bacterial infection or uncontrolled systemic fungal infection;
* - c.Diabetes that cannot be controlled by combination therapy;
* - d.Severe cardiac disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (NYHA [NYHA] class III or higher), and severe arrhythmia;
* - e.Patients with hypertension that cannot be controlled by drug therapy, that is, those with hypertension who cannot be reduced to the following range after combined treatment with 2 drugs (systolic blood pressure <160 mmHg, diastolic blood pressure <100 mmHg);
* - f.Comorbid psychiatric or psychotic disorders or central nervous system disorders;
* 12.receiving other interventional clinical trial medications within 1 month prior to signing the Informed Consent Form (ICF);
* 13.Pregnant or breastfeeding women, women/men of chil - dbearing age who have a plan to become pregnant during the trial period and within 6 months after the end of the trial;
* 14.Patients with a history of severe allergic reaction, or allergic reaction to any drug and related excipient specified in the protocol and judged by the investigator not suitable for enrollment;
* 15.Other conditions that the investigator considers unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT). | Day 0~ 28 after treatment with CG-105-12 injection（D0）
Adverse event related laboratory tests, vital signs, physical examination | Up to 12 months after treatment with CG-105-12 injection

SECONDARY OUTCOMES:
Objective response rate (ORR); | Up to 12 months following CG-105-12 injection
  Proportion of subjects with multiple myeloma receiving response(sCR,CR, VGPR or PR) after treatment with CG-105-12 injection
Duration of remission (DOR) after administration; | Up to 12 months following CG-105-12 injection
  Time from the first assessment of PR and above for multiple myeloma to the first assessment of disease progression or death from any cause
Progression free survival (PFS); | Up to 12 months after treatment with CG-105-12 injection
  Time from the beginning of treatment with CG-105-12 to the first disease progression or death from any cause
Overall survival (OS) | Up to 15 years
  Time from receiving CG-105-12 treatment(Day0) to death (for any reason)
Time to remission (TTR) | Up to 12 months after treatment with CG-105-12 injection
  Time interval from receiving CG-105-12 treatment（Day 0） to first recording to disease remission
Time to complete remission (TTCR): | Up to 12 months following CG-105-12 injection
  The time interval between the subject receiving CG-105-12 treatment（Day 0） and the first recorded complete remission of the disease
MRD efficacy evaluation | Up to 12 months following CG-105-12 injection
  Flow MRD evaluation, including MRD negative proportion and MRD negative duration
CG-105-12 cell count | Up to 12 months following CG-105-12 injection
  Pharmacokinetic (PK) parameters (including but not limited to Cmax, AUC, Tmax, tlast, etc.) were used to detect the concentration of CG-105-12 cells.
The transgenic level of CG-105-12. | Up to 12 months following CG-105-12 injection
  Pharmacokinetic (PK) parameters (including but not limited to Cmax, AUC, Tmax, tlast, etc.) were used to detect the transgenic level of CG-105-12.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, Study Director — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided